CLINICAL TRIAL: NCT06345729
Title: A Phase 3, Randomized, Double-blind, Multicenter Study of MK-1084 in Combination With Pembrolizumab Compared With Pembrolizumab Plus Placebo as Firstline Treatment of Participants With KRAS G12C-Mutant, Locally Advanced or Metastatic NSCLC With PD-L1 TPS ≥50% (KANDLELIT-004)
Brief Title: A Study of Calderasib (MK-1084) Plus Pembrolizumab (MK-3475) in Participants With KRAS G12C Mutant Non-small Cell Lung Cancer (NSCLC) With Programmed Cell Death Ligand 1 (PD-L1) Tumor Proportion Score (TPS) ≥50% (MK-1084-004/KANDLELIT-004)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1084-004; MK-1084-004 (Other: MSD); U1111-1296-8093 (Registry Identifier: UTN); 2023-507776-42-00 (Registry Identifier: EU CT); jRCT2031240213 (Registry Identifier: jRCT); PHRR241128-007796 (Registry Identifier: PHRR); KANDLELIT-004 (Other: MSD)
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2); Kirsten rat sarcoma viral oncogene homolog G12C (KRAS G12C)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Calderasib with Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles and calderasib by oral tablets until discontinuation criterion is met.
  Interventions: Drug: Calderasib; Biological: Pembrolizumab
- Placebo with Pembrolizumab (Active Comparator): Participants receive pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles and placebo by oral tablets once daily until discontinuation criterion is met.
  Interventions: Other: Placebo; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Calderasib — Oral tablets
  Other Names: MK-1084
  Arms: Calderasib with Pembrolizumab
Other: Placebo — Oral tablets
  Arms: Placebo with Pembrolizumab
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA ®

SUMMARY:
This is a study evaluating the efficacy and safety of calderasib with pembrolizumab as first-line treatment in participants with locally advanced or metastatic non-small cell lung cancer (NSCLC) with identified Kirsten rat sarcoma viral oncogene homolog G12C (KRAS G12C) mutation and programmed cell death ligand 1 (PD-L1) tumor proportion score (TPS) ≥50%. There are two primary study hypotheses:

Hypothesis 1: Combination of calderasib and pembrolizumab is superior to placebo plus pembrolizumab with respect to progression free survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by blinded independent central review (BICR).

Hypothesis 2: Combination of calderasib plus pembrolizumab is superior to placebo plus pembrolizumab with respect to overall survival (OS).

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC)
* Has newly diagnosed Stage IIIB/IIIC NSCLC, not eligible for curative resection or curative chemotherapy/radiation as determined by a multidisciplinary tumor board and/or by radiation oncologist, surgeon, and medical oncologist or Stage IV (M1a, M1b, or M1c) by American Joint Committee on Cancer (AJCC) Staging Manual, Version 8
* Provides an archival tumor tissue sample (≤5 years) or newly obtained core, incisional, or excisional biopsy of a tumor lesion not previously irradiated to enable central laboratory testing of kirsten rat sarcoma (KRAS) G12C mutation status, PD-L1 status, and biomarker research
* If have had adverse events (AEs) due to previous anticancer therapies, must have recovered to < Grade 1 or baseline
* If human immunodeficiency virus (HIV)-infected, must have well controlled HIV on antiretroviral therapy (ART)
* If Hepatitis B surface antigen (HBsAg) positive, have received Hepatitis B Virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load
* If a participant has a history of Hepatitis C virus (HCV) infection, HCV viral load is undetectable

Exclusion Criteria:

* Has diagnosis of small cell lung cancer. For mixed tumors, if small cell elements are present, the participant is ineligible
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous clear history of inflammatory bowel disease
* Has known history of, or active, neurologic paraneoplastic syndrome
* Has an active infection requiring systemic therapy, with exceptions
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease
* Has one or more of the following ophthalmological findings/conditions: intraocular pressure >21 mmHg and/or any diagnosis of glaucoma, diagnosis of central serous retinopathy, retinal vein occlusion, or retinal artery occlusion, diagnosis of retinal degenerative disease
* Has received prior systemic anticancer therapy for their locally advanced or metastatic NSCLC
* Has received radiation therapy to the lung that is >30 Gray within 6 months of start of study intervention
* Has received radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not required corticosteroids, and not have had radiation pneumonitis
* Has known active central nervous system metastases and/or carcinomatous meningitis
* Known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Has history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Is HIV-infected and has a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has history of allogenic tissue/solid organ transplant
* Has not fully recovered from any effects of major surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2029-02-19 (Estimated); Study Completion 2031-02-18 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 42 months
  PFS is defined as the time from randomization until either documented disease progression per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) or death due to any cause, whichever occurs first. PFS as determined by blinded independent central review (BICR) will be presented.
Overall Survival (OS) | Up to approximately 56 months
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 42 months
  ORR is defined as the percentage of participants with Complete Response or Partial Response per RECIST1.1. The percentage of participants who experience CR or PR as assessed by BICR will be presented.
Duration of Response (DOR) | Up to approximately 42 months
  For participants who demonstrate confirmed CR or PR per RECIST 1.1 as assessed by BICR, duration of response is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Number of Participants Who Experience One or More Adverse Event (AEs) | Up to approximately 56 months
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who experience an AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an Adverse Event (AE) | Up to approximately 56 months
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who discontinue study treatment due to an AE will be presented.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score | Baseline and Up to approximately 24 months
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in the score of EORTC QLQ-C30 Items 29 and 30 will be presented. Higher scores indicate a better overall health status.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Physical Functioning (Items 1-5) Score | Baseline and Up to approximately 24 months
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). The change from baseline in the score of EORTC QLQ-C30 Items 1-5 will be presented. Higher scores indicate a better level of functioning.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Role Functioning (Items 6 and 7) Score | Baseline and Up to approximately 24 months
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 2 questions about their role functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). The change from baseline in the score of EORTC QLQ-C30 Items 6-7 will be presented. Higher scores indicate a better level of functioning.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Dyspnea (Item 8) Score | Baseline and Up to approximately 24 months
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). The change from baseline in the score of EORTC QLQ-C30 Item 8 will be presented. A higher score indicates a worse level of dyspnea.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Lung Cancer-Specific Questionnaire Module (EORTC QLQ-C13) Cough (Item 31) Score | Baseline and Up to approximately 24 months
  The EORTC QLQ-C13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant response to the question "Have you coughed?" is scored on a 4-point scale (1=Not at All to 4=Very Much). The change from baseline in the score of EORTC QLQ-C13 Item 31 will be presented. A higher score indicates more frequent coughing.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Lung Cancer-Specific Questionnaire Module (EORTC QLQ-LC13) Chest pain (Item 40) Score | Baseline and Up to approximately 24 months
  The EORTC QLQ-C13 is lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant response to the question "Have you had pain in your chest?" is scored on a 4-point scale (1=Not at All to 4=Very Much). The change from baseline in the score of EORTC QLQ-C13 Item 40 will be presented. A higher score indicates a worse level of chest pain.
Time to Deterioration (TTD) in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score | Baseline and Up to approximately 24 months
  TTD is defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) from baseline in global health status (GHS) and quality of life (QoL) (EORTC QLQ-C30 Items 29 and 30) score. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10 point negative change (decrease) from baseline in GHS and QoL, will be presented. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Physical Functioning (Items 1-5) Score | Baseline and Up to approximately 24 months
  TTD is defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) from baseline in physical functioning (EORTC QLQ-C30 Items 1-5) score. The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10 point negative change (decrease) from baseline in physical functioning score, will be presented. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Role Functioning (Items 6 and 7) Score | Baseline and Up to approximately 24 months
  TTD is defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) from baseline in role functioning (EORTC QLQ-C30 Items 6 and 7) score. The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 2 questions about their role functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10 point negative change (decrease) from baseline in role functioning score, will be presented. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Dyspnea (Item 8) Score | Baseline and Up to approximately 24 months
  TTD is defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) from baseline in dyspnea (EORTC QLQ-C30 Item 8) score. The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10 point negative change (decrease) from baseline in dyspnea score, will be presented. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in European Organization for Research and Treatment of Cancer Quality of Life Lung Cancer-Specific Questionnaire Module (EORTC QLQ-C13) Cough (Item 31) Score | Baseline and Up to approximately 24 months
  TTD is defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) from baseline in cough (EORTC QLQ-C13 Item 31) score. The EORTC QLQ-C13 is lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant response to the question "Have you coughed?" is scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10 point negative change (decrease) from baseline in cough score, will be presented. A longer TTD indicates a better outcome.
Time to Deterioration (TTD) in European Organization for Research and Treatment of Cancer Quality of Life Lung Cancer-Specific Questionnaire Module (EORTC QLQ-C13) Chest pain (Item 40) Score | Baseline and Up to approximately 24 months
  TTD is defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) from baseline in chest pain (EORTC QLQ-C13 Item 40) score. The EORTC QLQ-C13 is lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant response to the question "Have you had pain in your chest?" is scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10 point negative change (decrease) from baseline chest pain score, will be presented. A longer TTD indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (207):
- United States (15):
  - CBCC Global Research, Inc. ( Site 0123), Bakersfield, California
  - Beverly Hills Cancer Center ( Site 0116), Beverly Hills, California
  - Stamford Hospital ( Site 0136), Stamford, Connecticut
  - Mount Sinai Cancer Center ( Site 0137), Miami Beach, Florida
  - Orchard Healthcare Research Inc. ( Site 0115), Skokie, Illinois
  - Truman Medical Center ( Site 0126), Kansas City, Missouri
  - Cox Medical Center North ( Site 0133), Springfield, Missouri
  - St. Vincent Frontier Cancer Center-Research ( Site 0105), Billings, Montana
  - Atlantic Health System Morristown Medical Center ( Site 0121), Morristown, New Jersey
  - New York Oncology Hematology, P.C. ( Site 0132), Albany, New York
  - University of Cincinnati Medical Center-University of Cincinnati Cancer Center ( Site 0103), Cincinnati, Ohio
  - Kettering Health Main Campus-Kettering Health Cancer Center ( Site 0106), Kettering, Ohio
  - Lancaster General Hospital - Ann B Barshinger Cancer Institute ( Site 0134), Lancaster, Pennsylvania
  - Oncology Consultants P.A. ( Site 0113), Houston, Texas
  - Circuit Clinical/SSM Health Dean Medical Group ( Site 0129), Madison, Wisconsin
- Argentina (5):
  - AUSTRAL MEDICAL CENTER ( Site 0302), CABA, Buenos Aires
  - Centro Oncologico Korben ( Site 0304), CABA, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0300), Mar del Plata, Buenos Aires
  - Fundacion Estudios Clinicos ( Site 0306), Rosario, Santa Fe Province
  - Sanatorio Parque ( Site 0301), Rosario, Santa Fe Province
- Australia (3):
  - Chris O'Brien Lifehouse ( Site 3000), Camperdown, New South Wales
  - Frankston Hospital ( Site 3002), Frankston, Victoria
  - One Clinical Research ( Site 3001), Nedlands, Western Australia
- Austria (2):
  - Medizinische Universität Graz-Klinische Abteilung für Pulmonologie ( Site 2401), Graz, Styria
  - Klinik Floridsdorf-Abteilung für Innere Medizin und Pneumologie ( Site 2400), Vienna
- Brazil (10):
  - Hospital Mario Penna ( Site 0436), Belo Horizonte, Minas Gerais
  - Hospital de Câncer de Recife ( Site 0447), Recife, Pernambuco
  - Oncoclínica Oncologistas Associados ( Site 0441), Teresina, Piauí
  - Liga Norte Riograndense Contra o Câncer ( Site 0439), Natal, Rio Grande do Norte
  - Hospital de Caridade de Ijuí ( Site 0438), Ijuí, Rio Grande do Sul
  - Hospital de Clínicas de Passo Fundo ( Site 0442), Passo Fundo, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre-Centro Multidisciplinar de Pesquisa Clínica ( Site 0435), Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos-Unidade de Pesquisa Clínica ( Site 0437), Barretos, São Paulo
  - Instituto Nacional de Câncer - INCA ( Site 0446), Rio de Janeiro
  - Americas ( Site 0431), Rio de Janeiro
- Bulgaria (3):
  - MBAL Uni Hospital-Department of Medical Oncology ( Site 1000), Panagyurishte, Pazardzhik
  - Multiprofile Hospital for Active Treatment SerdikaМЕD EOOD-Second Department of Medical Oncology ( Site 1002), Sofia, Sofia (stolitsa)
  - MHAT - Heart and Brain ( Site 1006), Pleven
- Canada (6):
  - CancerCare Manitoba ( Site 0210), Winnipeg, Manitoba
  - QEII Health Sciences Centre - Victoria General Site-Dept. of Medical Oncology ( Site 0208), Halifax, Nova Scotia
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0205), Hamilton, Ontario
  - Sunnybrook Research Institute ( Site 0206), Toronto, Ontario
  - St. Marys Hospital Center ( Site 0204), Montreal, Quebec
  - Centre integre universitaire de sante et de services sociaux de la Mauricie-et-du-centre-du-quebec ( Site 0207), Trois-Rivières, Quebec
- Chile (5):
  - Clinica Universidad Catolica del Maule-Oncology ( Site 0500), Talca, Maule Region
  - Orlandi Oncologia-Oncology ( Site 0503), Santiago, Region M. de Santiago
  - FALP-UIDO ( Site 0501), Santiago, Region M. de Santiago
  - Centro de Oncología de Precisión-Oncology ( Site 0502), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0504), Santiago, Region M. de Santiago
- China (45):
  - Anhui Provincial Cancer Hospital ( Site 3136), Hefei, Anhui
  - Beijing Cancer hospital ( Site 3133), Beijing, Beijing Municipality
  - Beijing Cancer hospital ( Site 3134), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital-pneumology department ( Site 3102), Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University ( Site 3104), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital ( Site 3119), Chongqing, Chongqing Municipality
  - Army Medical Center of People's Liberation Army ( Site 3142), Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital ( Site 3127), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University ( Site 3148), Xiamen, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 3108), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 3128), Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center ( Site 3137), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital ( Site 3123), Harbin, Heilongjiang
  - JIAMUSI TUBERCULOSIS HOSPITAL(CANCER HOSPITAL) ( Site 3124), Jiamusi, Heilongjiang
  - Henan Cancer Hospital ( Site 3149), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 3113), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 3126), Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University ( Site 3130), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 3141), Changsha, Hunan
  - Nanjing Gulou Hospital ( Site 3122), Nanjing, Jiangsu
  - Nanjing First Hospital ( Site 3154), Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University ( Site 3146), Suzhou, Jiangsu
  - Affiliated Hospital of Jiangnan University(Wuxi Fourth People's Hospital ) ( Site 3155), Wuxi, Jiangsu
  - The Second Affiliated Hospital of Nanchang University ( Site 3139), Nanchang, Jiangxi
  - The First affiliated hospital of Nanchang University (Xianghu campus) ( Site 3138), Nanchang, Jiangxi
  - Jilin Province Tumor Hospital ( Site 3107), Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University ( Site 3150), Xi'an, Shaanxi
  - Shandong Cancer Hospital ( Site 3116), Jinan, Shandong
  - LinYi Cancer Hospital ( Site 3111), Linyi, Shandong
  - Shanghai Chest Hospital ( Site 3100), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center ( Site 3144), Shanghai, Shanghai Municipality
  - Zhongshan Hospital,Fudan University ( Site 3143), Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital ( Site 3131), Taiyuan, Shanxi
  - The Second Affiliated Hospital of Air Force Medical University ( Site 3117), Xian, Shanxi
  - The Second Affiliated Hospital of Air Force Medical University ( Site 3152), Xian, Shanxi
  - The Third People's Hospital of Chengdu (CDTPH) ( Site 3157), Chengdu, Sichuan
  - West China Hospital, Sichuan University ( Site 3140), Chengdu, Sichuan
  - Sichuan Cancer hospital. ( Site 3109), Chengdu, Sichuan
  - The Second People's Hospital of Neijiang ( Site 3105), Neijiang, Sichuan
  - Xinjiang Medical University Cancer Hospital - Urumqi ( Site 3101), Ürümqi, Xinjiang
  - Yunnan Province Cancer Hospital ( Site 3153), Kunming, Yunnan
  - The first Affiliated Hospital, Zhejiang University School of Medicine ( Site 3115), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine ( Site 3121), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 3145), Linhai, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 3151), Wenzhou, Zhejiang
- France (6):
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand ( Site 1103), Dijon, Bourgogne-Franche-Comté
  - Centre Hospitalier Universitaire de Nîmes - Institut de Cancérologie du Gard - Hôpital Universitaire ( Site 1106), Nîmes, Gard
  - Clinique Teissier Groupe ( Site 1100), Valenciennes, Nord
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne-ONCOLOGY ( Site 1101), Clermont-Ferrand, Puy-de-Dome
  - Centre Hospitalier d'Avignon-Service d'Oncologie médicale et d'hématologie clinique ( Site 1104), Avignon, Vaucluse
  - Hôpital Ambroise Paré-Department of Respiratory Diseases and Thoracic Oncology ( Site 1105), Boulogne-Billancourt, Île-de-France Region
- Georgia (8):
  - High Technology Hospital Medcenter ( Site 1203), Batumi, Adjara
  - Caucasus Medical Centre ( Site 1202), Tbilisi, Adjara
  - American Hospital Network LLC ( Site 1208), Tbilisi
  - Todua Clinic, LLC ( Site 1204), Tbilisi
  - TSMU and Ingorokva High Medical Technology University Clinic LTD ( Site 1201), Tbilisi
  - New Hospitals ( Site 1200), Tbilisi
  - Cancer Research Centre. Mardaleishvili Medical Centre ( Site 1205), Tbilisi
  - Tbilisi Institute of Medicine ( Site 1206), Tbilisi
- Germany (2):
  - Marienhospital Stuttgart ( Site 1302), Stuttgart, Baden-Wurttemberg
  - Krankenhaus Bethanien ( Site 1303), Solingen, North Rhine-Westphalia
- Greece (5):
  - UNIVERSITY HOSPITAL OF PATRAS-DIVISION OF ONCOLOGY ( Site 1402), Pátrai, Achaia
  - THORACIC GENERAL HOSPITAL OF ATHENS "I SOTIRIA"-3rd Dept of Internal Medicine and Laboratory, Oncol ( Site 1400), Athens, Attica
  - University General Hospital of Larissa-Oncology Clinic ( Site 1403), Larissa, Thessaly
  - Agios Loukas Clinic ( Site 1404), Thessaloniki
  - G. Papanikolaou General Hospital-Pulmonary Clinic of Aristotle University of Thessaloniki ( Site 1405), Thessaloniki
- Sir H. N. Reliance Foundation Hospital and Research Centre ( Site 3201), Mumbai, Maharashtra, India
- Italy (10):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-Oncologia clinica sperimentale Toraco-Polmonare ( Site 1607), Napoli, Campania
  - Ospedale Santa Maria delle Croci ( Site 1606), Ravenna, Emilia-Romagna
  - CRO-IRCCS-Clinical Oncology ( Site 1605), Aviano, Friuli Venezia Giulia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -Medical Oncology ( Site 1601), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1600), Milan, Lombardy
  - Istituto Europeo di Oncologia IRCCS-Divisione di Oncologia Toracica ( Site 1604), Milan, Lombardy
  - A.O.R.N. Ospedale dei Colli - Monaldi V.-U.O.C Pneumologia Oncologica DH PNL ONC ( Site 1602), Naples, Napoli
  - Istituto Nazionale Tumori Regina Elena-Oncologia Medica 2 ( Site 1609), Rome, Roma
  - Azienda USL Toscana Nord Ovest_Ospedale Civile di Livorno-UOC Oncologia Medica Livorno ( Site 1608), Livorno, Tuscany
  - IOV - Istituto Oncologico Veneto IRCCS UOSD - Unità di ricerca clinica ( Site 1603), Padua
- Japan (25):
  - Nagoya University Hospital ( Site 3309), Nagoya, Aichi-ken
  - Fujita Health University Hospital ( Site 3310), Toyoake, Aichi-ken
  - National Cancer Center Hospital East ( Site 3303), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 3315), Matsuyam, Ehime
  - National Hospital Organization Kyushu Cancer Center ( Site 3316), Fukuoka, Fukuoka
  - Kurume University Hospital ( Site 3317), Kurume, Fukuoka
  - Gunma Prefectural Cancer Center ( Site 3302), Ōta, Gunma
  - Sapporo Medical University Hospital ( Site 3324), Sapporo, Hokkaido
  - Kanazawa University Hospital ( Site 3308), Kanazawa, Ishikawa-ken
  - St. Marianna University Hospital ( Site 3320), Kawasaki, Kanagawa
  - Matsusaka Municipal Hospital ( Site 3311), Matsusaka, Mie-ken
  - Miyagi Cancer Center ( Site 3301), Natori-shi, Miyagi
  - Sendai Kousei Hospital ( Site 3300), Sendai, Miyagi
  - Kansai Medical University Hospital ( Site 3312), Hirakata, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 3313), Takatsuki, Osaka
  - Saitama Prefectural Cancer Center ( Site 3304), Kitaadachi-gun, Saitama
  - Nippon Medical School Hospital ( Site 3306), Bunkyo, Tokyo
  - Toho University Omori Medical Center ( Site 3319), Ōta-ku, Tokyo
  - Tokyo Medical University Hospital ( Site 3307), Shinjuku, Tokyo
  - National Center for Global Health and Medicine ( Site 3305), Shinjuku, Tokyo
  - Chiba University Hospital ( Site 3322), Chiba
  - Hiroshima City Hiroshima Citizens Hospital ( Site 3314), Hiroshima
  - Saiseikai Kumamoto Hospital ( Site 3318), Kumamoto
  - Niigata University Medical & Dental Hospital ( Site 3323), Niigata
  - Osaka Metropolitan University Hospital ( Site 3321), Osaka
- Mexico (3):
  - Arké SMO S.A. de C.V. ( Site 0602), Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Hematologia and Oncologia ( Site 0600), Monterrey, Nuevo León
  - Oaxaca Site Management Organization S.C. ( Site 0603), Oaxaca City
- Netherlands (4):
  - Ziekenhuis Gelderse Vallei ( Site 1705), Ede, Gelderland
  - Ziekenhuis St. Jansdal-Poli Longziekten ( Site 1701), Harderwijk, Gelderland
  - Isala, locatie Zwolle-Poli Longziekten ( Site 1700), Zwolle, Overijssel
  - Universitair Medisch Centrum Utrecht ( Site 1704), Utrecht
- Auckland City Hospital ( Site 3400), Auckland, New Zealand
- Philippines (4):
  - The Medical City ( Site 3507), Pasig, National Capital Region
  - Lung Center of the Philippines-Pulmonary, Critical Care and Sleep Medicine ( Site 3503), Quezon City, National Capital Region
  - Veterans Memorial Medical Center-Section of Oncology ( Site 3505), Quezon City, National Capital Region
  - ST. LUKE'S MEDICAL CENTER-Medical oncology ( Site 3501), Quezon City, National Capital Region
- Poland (5):
  - Szpital Specjalistyczny im. Henryka Klimontowicza ( Site 1801), Gorlice, Lesser Poland Voivodeship
  - Pratia MCM Krakow ( Site 1808), Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny nr 4 w Lublinie ( Site 1805), Lublin, Lublin Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 1800), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 1804), Przemyśl, Podkarpackie Voivodeship
- Romania (6):
  - Centrul de Diagnostic si Tratament Provita. ( Site 1992), Bucharest, București
  - Centrul de Oncologie Sfantul Nectarie-Medical ( Site 1994), Craiova, Dolj
  - Cabinet Medical Oncomed ( Site 1998), Timișoara, Timiș County
  - SC ONCO CARD SRL ( Site 1995), Brasov
  - Institutul Oncologic Cluj-Oncologie Medicala ( Site 1999), Cluj-Napoca
  - Sigmedical Services SRL ( Site 1997), Suceava
- South Korea (7):
  - The Catholic University of Korea, Incheon St. Mary's Hospital ( Site 3606), Bupyeong-gu, Incheon
  - Chonnam National University Hwasun Hospital-Pulmonology ( Site 3604), Hwasun, Jeonranamdo
  - The Catholic University Of Korea St. Vincent's Hospital-Medical Oncology ( Site 3600), Suwon, Kyonggi-do
  - Pusan National University Yangsan Hospital-Lung Cancer Clinic ( Site 3603), Yangsan, Kyongsangnam-do
  - Chungnam national university hospital ( Site 3602), Junggu, Taejon-Kwangyokshi
  - Kyung Hee University Hospital ( Site 3605), Seoul
  - Korea University Guro Hospital ( Site 3601), Seoul
- Spain (6):
  - Hospital Insular de Gran Canaria-Oncology ( Site 2019), Las Palmas de Gran Canaria, Las Palmas
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON-ONCOLOGY ( Site 2012), Madrid, Madrid, Comunidad de
  - H.R.U Málaga - Hospital General-Oncology ( Site 2014), Málaga, Malaga
  - Hospital Universitari Vall d Hebron ( Site 2010), Barcelona
  - Hospital Universitario Fundación Jiménez Díaz-Oncology & Hematology ( Site 2017), Madrid
  - Hospital Universitario Virgen Macarena-Unidad de Investigación Oncológica ( Site 2015), Seville
- Turkey (Türkiye) (8):
  - Ege Universitesi Hastanesi-Chest Diseases Department ( Site 2102), Bornova, İzmir
  - Adana Medical Park Seyhan Hastanesi-Medikal Onkoloji ( Site 2107), Adana
  - SBU GULHANE EGITIM VE ARASTIRMA HASTANESI Onkoloji ( Site 2104), Ankara
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 2101), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 2106), Ankara
  - Ankara Bilkent Şehir Hastanesi ( Site 2100), Ankara
  - Medipol Mega Universite Hastanesi-oncology ( Site 2105), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 2103), Istanbul
- Ukraine (10):
  - COMMUNAL NONPROFIT ENTERPRISE "CLINICAL CENTER OF ONCOLOGY, HEMATOLOGY, TRANSPLANTOLOGY AND PALLIATI ( Site 2209), Cherkasy, Cherkasy Oblast
  - Regional Municipal Non-profit Enterprise "Bukovinian Clinica-structural unit of the clinical trials ( Site 2210), Chernivtsi, Chernivetska Oblast
  - Medical Center "Mriya Med-Service"-Clinical Research Department ( Site 2215), Kryvyi Rih, Dnipropetrovsk Oblast
  - Communal Non-Commercial Enterprise "Prykarpatski Clinical On-Surgery department #2 ( Site 2202), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Kirovohrad Regional Oncology Center-Chemotherapy department ( Site 2204), Kropyvnytskyi, Kirovohrad Oblast
  - Medical Center "MedOffice Group" ( Site 2219), Kiev, Kyivska Oblast
  - Rivne Regional Clinical Hospital ( Site 2205), Rivne, Rivne Oblast
  - ME RIVNE REGIONAL ANTITUMOR CENTER ( Site 2920), Rivne, Rivne Oblast
  - Communal Noncommercial Enterprise "Podillia Regional Oncolog-Cardiothoracic department ( Site 2211), Vinnytsia, Vinnytsia Oblast
  - ME Volyn Regional Clinical Hospital of the Volyn Regional Council ( Site 2216), Lutsk, Volyn Oblast
- United Kingdom (2):
  - Milton Keynes Hospital ( Site 2304), Milton Keynes, Buckinghamshire
  - Royal Devon & Exeter Hospital-Oncology ( Site 2302), Exeter, Devon

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26314&tenant=MT_MSD_9011